CLINICAL TRIAL: NCT00574678
Title: ACT: Analyzing the Composition of Tears to Identify Cancer (Breast, Ovarian, Colon)
Brief Title: Analyzing the Composition of Tears to Identify Cancer
Acronym: ACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Tenenbaum Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 71853
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2016-02

CONDITIONS: Breast Cancer; Ovarian Cancer; Colon Cancer; Benign Disease
Keywords: Screening tool for cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms | interventions — Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention)
  Interventions: Other: Tear collection

INTERVENTIONS:
Other: Tear collection — A tear sample (~75 microliters in a tuberculin syringe with the needle removed) will be taken at time of the initial clinic visit. After collection, the tears will be put directly on ice and taken to the lab. If it is not possible to obtain natural tears, an "eye wash" method using sterile saline will be employed and the fluid collected using the aforementioned technique. The SELDI-MS process will be conducted on the specimen immediately. The remainder of the tear specimen will be stored in a -80ºC freezer until completely analyzed.
  Other Names: SELDI-MS

SUMMARY:
This study will further evaluate the use of protein identification or protein pattern (signature) found in tears. We hypothesize that differences exist between the protein profile in tear fluid from patients with versus without cancer.

DETAILED DESCRIPTION:
Specifically, this study will compare the protein profile in tear fluid from patients with breast, ovarian or colon cancer versus "normal male and female patients" for differences that show promise as a diagnostic indicator. If such differences can be found, then their diagnostic potential will be assessed and developed further in a subsequent study. The long-term goal of this project will be to develop a screening tool for the detection of breast and/or other cancers.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18-100 years old
* Patients who present for a routine check-up
* Patients who present for the evaluation of an abnormal exam or test (mammogram, ultrasound, MRI, PET, etc.)
* May or may not have a mass present
* Patients who present for the evaluation of a palpable lump or mass
* Patients may be pre or post biopsy for a mass, as long as there is a portion of the mass remaining

Exclusion Criteria:

* Patient < 18 y/o or > 100 y/o
* Concurrent eye infection or trauma
* Active conjunctivitis
* Abnormal production of tears (too much or too little)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
This study will further evaluate the use of tumor markers (substances in body fluids that may be elevated as a consequence of certain diseases or conditions) in the diagnosis of breast and/or other cancers. | Collection of specimen and analysis with SELDI-MS

CONTACTS AND LOCATIONS:
Overall Officials: V. Suzanne Klimberg, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States